CLINICAL TRIAL: NCT01752868
Title: Can Fish Oil and Phytochemical Supplements Mimic Anti-Aging Effects of Calorie Restriction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJH 6936-33
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Dietary Supplements

ARMS (2):
- supplement (Experimental)
  Interventions: Dietary Supplement: Supplement
- control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Supplement — Participants in this group will take the following nutritional supplements on a daily basis: curcumin, fish oil, resveratrol, sesamin, Acetyl-L-carnitine, lipoic acid, green and black teas, quercetin, pomegranate, cinnamon bark.
  Arms: supplement

SUMMARY:
The purpose of this study is to determine if a combination of 10 nutritional supplements provide health benefits that are consistent with protection against age-related disease. All supplements have been shown in previous studies to have health benefits when administered alone. The hypothesis is that 6 months of taking 10 nutritional supplements each day will provide beneficial changes in healthy related measures.

ELIGIBILITY:
Inclusion Criteria:

* age 40-60 yr
* body mass index of 21 - 30 kg/m2
* sedentary to moderately active
* eating a typical US diet

Exclusion Criteria:

* history of any chronic disease other than mild osteoarthritis
* use of medications other than occasional use of non-steroidal anti-inflammatory drugs, antihistamines, antacids or laxatives
* use of nutritional supplements
* smoking
* alcohol intake greater than two drinks per day for women and three drinks per day for men

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral pulse wave velocity | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fontana, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States